CLINICAL TRIAL: NCT07223775
Title: Kangaroo Care in the Operating Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00148361
Record Dates: First submitted 2025-10-10; First posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Cesarean Section; Skin to Skin; Kangaroo Care
MeSH Terms: interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kangaroo Care (Experimental): This group received immediate post delivery via Cesarean section skin-to-skin interaction.
  Interventions: Procedure: Kangaroo Care
- Standard OR care (No Intervention): This group received standard care post delivery via Cesarean section.

INTERVENTIONS:
Procedure: Kangaroo Care — Patients undergoing a planned cesarean section and assigned to the intervention group would get to hold their infant skin to skin immediately after delivery.
  Arms: Kangaroo Care

SUMMARY:
The study was done to learn how kangaroo care in the operating room help mothers and infants.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Scheduled Cesarean Sections at KUMC
* Term delivery

Exclusion Criteria:

* Priority, urgent and emergent Cesarean sections
* Planned general anesthesia
* Fetal anomalies
* Fetal aneuploidy/genetic syndrome
* Abnormal fetal dopplers
* Placental previa/accreta
* Multiple gestations
* Preeclampsia with severe features

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Maternal C-section satisfaction | Delivery
  Assess maternal satisfaction using Likert-scale surveys (like very satisfied...very unsatisfied)
Maternal pain level | Delivery
  Assess maternal pain using Likert-scale surveys (like no pain...unbearable pain)
Maternal pain medication needed | Delivery
  Assess maternal pain medications given before, during and after cesarean section delivery from the patients' chart
Cesarean section blood loss | Delivery
  Assess quantitative blood loss (QBL) of the cesarean section from the patients' chart
Neonatal morbidity | Delivery
  Assess neonatal morbidity by collecting neonatal APGAR scores from the patients' chart
Neonatal morbidity | Delivery
  Assess neonatal morbidity by collecting skin to skin from the patients' chart
Neonatal morbidity | Delivery
  Assess neonatal morbidity by collecting neonatal ICU admissions rate from the patients' chart

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Gray, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States